CLINICAL TRIAL: NCT02765126
Title: Clifford Craig Vaccine Trial Centre: Heterologous Effect of Diptheria, Tetanus, Acellular Pertussis Vaccination on Influenza Vaccine Challenge in the Elderly
Brief Title: Heterologous Effect of Diptheria, Tetanus, Acellular Pertussis Vaccination on Influenza Challenge in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clifford Craig Medical Research Trust (Other)
Collaborators: Monash University (Other); The Peter Doherty Institute for Infection and Immunity (Other); University of Sao Paulo (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H0015460
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Heterologous Effects of Vaccines
MeSH Terms: interventions — Influenza Vaccines; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Diphtheria-tetanus-acellular pertussis vaccine administered day 0, followed by seasonal influenza vaccination four weeks later. Blood testing to occur day 0 (prior to vaccine administration), 24 hours, 1 week, 4 weeks, 4 weeks + 24 hours, 5 weeks, 8 weeks and 30 weeks. Stool samples to be taken at day 0 and 1 week post-vaccination.
  Interventions: Biological: Seasonal influenza vaccine; Biological: Diphtheria-tetanus-acellular pertussis vaccine
- Group 2 (Active Comparator): Seasonal influenza vaccine administered on day 0, to be offered DTP vaccine at week 26. Blood testing to occur day 0 (prior to vaccine administration), 24 hours, 1 week 1, 4 weeks and 26 weeks. Stool samples to be taken at day 0 and 1 week post-vaccination.
  Interventions: Biological: Seasonal influenza vaccine; Biological: Diphtheria-tetanus-acellular pertussis vaccine
- Group 3 (Active Comparator): Seasonal influenza vaccine and DTP vaccine administered together on day 0. Blood testing to occur day 0 (prior to vaccine administration), 24 hours, 1 week 1, 4 weeks and 26 weeks. Stool samples to be taken at day 0 and 1 week post-vaccination.
  Interventions: Biological: Seasonal influenza vaccine; Biological: Diphtheria-tetanus-acellular pertussis vaccine

INTERVENTIONS:
Biological: Seasonal influenza vaccine — Intramuscular standard seasonal influenza vaccine
  Other Names: Quadrivalent Influenza Vaccine
Biological: Diphtheria-tetanus-acellular pertussis vaccine — Intramuscular DTaP vaccine
  Other Names: Boostrix vaccine

SUMMARY:
Vaccines can have non-targeted or heterologous (also called non-specific) immunological effects on the immune system i.e. effects other than inducing an immune response against the disease targeted by the vaccine. This trial aims to evaluate the non-specific immunological effects of two vaccines - diphtheria-tetanus-acellular pertussis (DTP) vaccine and seasonal influenza vaccine - in a cohort of elderly humans (>65 years of age) and healthy adult control subjects (30-50 years).

DETAILED DESCRIPTION:
This prospective randomised study aims to investigate the heterologous immunological effects of DTP and seasonal influenza (Flu) vaccination in an elderly Tasmanian population and healthy adults. The study will assess whether prior or concurrent administration of DTP with seasonal Flu vaccination affects generalised inflammation / immune homeostasis and gene expression, with a particular focus of inflammation reactive cells. It will also analyse for effects of DTP on the induction of vaccine-specific immunity to seasonal influenza vaccination (antibodies and cellular). Volunteers will be randomised to one of three vaccine groups and serial blood samples taken for immunological assays for up to 30 weeks.

The study is exploratory and will investigate vaccine effects on multiple immune parameters.

ELIGIBILITY:
Inclusion Criteria:

* Two study groups 30-50 years old >65 years old

Exclusion Criteria:

* Unwell on day of vaccination
* Temperature >38°C
* Active cancer
* Active autoimmune disease
* Diabetes mellitus
* Taking immunosuppressive drugs including steroids
* Any vaccination in last 3 months
* DT or DTaP vaccination in the last year
* Known allergy or contraindication to influenza or DTaP vaccination
* Pregnant or breastfeeding

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of inflammation reactive TNFR2+ regulatory T cells per mL of blood | 24 hours, 1 week, 4 weeks and 26 weeks
  Change over time in different vaccine groups of Tregs measured by flow cytometry.

SECONDARY OUTCOMES:
Whole human genome transcription profile by next generation sequencing in log2 expression levels | 24 hours
  Differential gene expression 24 hours after vaccination compared to baseline, and vaccine groups compared to see which genes / pathways are affected. Differential transcription determined for each gene, then analysed using modular analysis tools to determine vaccine effects.
Influenza-specific antibody titres to seasonal influenza vaccination | 4 weeks and 26 weeks
  Change over time in the different vaccine groups of titres measured by haemagglutination inhibition assay.
Pro-inflammatory (TNF) to anti-inflammatory (IL-10) cytokine ratio in stimulated blood in pg/mL | 24 hours, 1 week, 4 weeks and 26 weeks
  Change in TNF:IL-10 ratio post-vaccination over time as measured by cytokine multiplex assay of anti-CD3 stimulated PBMC.
Influenza-specific IFN-g CD4 T cell responses to seasonal influenza vaccination in pg/mL | 4 weeks and 26 weeks
  Change over time in the different vaccine groups of IFN-g levels in supernatants from CD4 T cells cultured with live influenza virus

CONTACTS AND LOCATIONS:
Overall Officials: Katie Flanagan, PhD FRACP, Principal Investigator — Clifford Craig Medical Research Trust
Locations (1):
- Clifford Craig Foundation, Launceston, Tasmania, Australia

IPD SHARING:
Plan to Share IPD: Yes
The transcriptome data will be de-identified and deposited in a pubic database. The de-identified microbiome data may well also be made publically available.

REFERENCES:
- [Background] Meeting of the Strategic Advisory Group of Experts on immunization, April 2014 -- conclusions and recommendations. Wkly Epidemiol Rec. 2014 May 23;89(21):221-36. No abstract available. English, French. PMID 24864348
- [Background] Aaby P, Martins CL, Garly ML, Bale C, Andersen A, Rodrigues A, Ravn H, Lisse IM, Benn CS, Whittle HC. Non-specific effects of standard measles vaccine at 4.5 and 9 months of age on childhood mortality: randomised controlled trial. BMJ. 2010 Nov 30;341:c6495. doi: 10.1136/bmj.c6495. PMID 21118875
- [Background] Sorup S, Benn CS, Poulsen A, Krause TG, Aaby P, Ravn H. Live vaccine against measles, mumps, and rubella and the risk of hospital admissions for nontargeted infections. JAMA. 2014 Feb 26;311(8):826-35. doi: 10.1001/jama.2014.470. PMID 24570246
- [Background] Aaby P, Benn C, Nielsen J, Lisse IM, Rodrigues A, Ravn H. Testing the hypothesis that diphtheria-tetanus-pertussis vaccine has negative non-specific and sex-differential effects on child survival in high-mortality countries. BMJ Open. 2012 May 22;2(3):e000707. doi: 10.1136/bmjopen-2011-000707. Print 2012. PMID 22619263
- [Background] Nichol KL, Nordin JD, Nelson DB, Mullooly JP, Hak E. Effectiveness of influenza vaccine in the community-dwelling elderly. N Engl J Med. 2007 Oct 4;357(14):1373-81. doi: 10.1056/NEJMoa070844. PMID 17914038
- [Background] Goodwin K, Viboud C, Simonsen L. Antibody response to influenza vaccination in the elderly: a quantitative review. Vaccine. 2006 Feb 20;24(8):1159-69. doi: 10.1016/j.vaccine.2005.08.105. Epub 2005 Sep 19. PMID 16213065
- [Background] Sasaki S, Sullivan M, Narvaez CF, Holmes TH, Furman D, Zheng NY, Nishtala M, Wrammert J, Smith K, James JA, Dekker CL, Davis MM, Wilson PC, Greenberg HB, He XS. Limited efficacy of inactivated influenza vaccine in elderly individuals is associated with decreased production of vaccine-specific antibodies. J Clin Invest. 2011 Aug;121(8):3109-19. doi: 10.1172/JCI57834. Epub 2011 Jul 25. PMID 21785218
- [Background] Grant EJ, Chen L, Quinones-Parra S, Pang K, Kedzierska K, Chen W. T-cell immunity to influenza A viruses. Crit Rev Immunol. 2014;34(1):15-39. doi: 10.1615/critrevimmunol.2013010019. PMID 24579700
- [Background] Saurwein-Teissl M, Lung TL, Marx F, Gschosser C, Asch E, Blasko I, Parson W, Bock G, Schonitzer D, Trannoy E, Grubeck-Loebenstein B. Lack of antibody production following immunization in old age: association with CD8(+)CD28(-) T cell clonal expansions and an imbalance in the production of Th1 and Th2 cytokines. J Immunol. 2002 Jun 1;168(11):5893-9. doi: 10.4049/jimmunol.168.11.5893. PMID 12023394
- [Background] Weston WM, Friedland LR, Wu X, Howe B. Vaccination of adults 65 years of age and older with tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine (Boostrix((R))): results of two randomized trials. Vaccine. 2012 Feb 21;30(9):1721-8. doi: 10.1016/j.vaccine.2011.12.055. Epub 2011 Dec 31. PMID 22212127
- [Background] Solana R, Tarazona R, Gayoso I, Lesur O, Dupuis G, Fulop T. Innate immunosenescence: effect of aging on cells and receptors of the innate immune system in humans. Semin Immunol. 2012 Oct;24(5):331-41. doi: 10.1016/j.smim.2012.04.008. Epub 2012 May 4. PMID 22560929
- [Background] Panda A, Qian F, Mohanty S, van Duin D, Newman FK, Zhang L, Chen S, Towle V, Belshe RB, Fikrig E, Allore HG, Montgomery RR, Shaw AC. Age-associated decrease in TLR function in primary human dendritic cells predicts influenza vaccine response. J Immunol. 2010 Mar 1;184(5):2518-27. doi: 10.4049/jimmunol.0901022. Epub 2010 Jan 25. PMID 20100933
- [Background] Baylis D, Bartlett DB, Syddall HE, Ntani G, Gale CR, Cooper C, Lord JM, Sayer AA. Immune-endocrine biomarkers as predictors of frailty and mortality: a 10-year longitudinal study in community-dwelling older people. Age (Dordr). 2013 Jun;35(3):963-71. doi: 10.1007/s11357-012-9396-8. Epub 2012 Mar 3. PMID 22388931
- [Background] Franceschi C, Capri M, Monti D, Giunta S, Olivieri F, Sevini F, Panourgia MP, Invidia L, Celani L, Scurti M, Cevenini E, Castellani GC, Salvioli S. Inflammaging and anti-inflammaging: a systemic perspective on aging and longevity emerged from studies in humans. Mech Ageing Dev. 2007 Jan;128(1):92-105. doi: 10.1016/j.mad.2006.11.016. Epub 2006 Nov 20. PMID 17116321
- [Background] Bruunsgaard H, Andersen-Ranberg K, Hjelmborg Jv, Pedersen BK, Jeune B. Elevated levels of tumor necrosis factor alpha and mortality in centenarians. Am J Med. 2003 Sep;115(4):278-83. doi: 10.1016/s0002-9343(03)00329-2. PMID 12967692
- [Background] Nikolich-Zugich J, Li G, Uhrlaub JL, Renkema KR, Smithey MJ. Age-related changes in CD8 T cell homeostasis and immunity to infection. Semin Immunol. 2012 Oct;24(5):356-64. doi: 10.1016/j.smim.2012.04.009. Epub 2012 May 1. PMID 22554418
- [Background] Ndure J, Flanagan KL. Targeting regulatory T cells to improve vaccine immunogenicity in early life. Front Microbiol. 2014 Sep 11;5:477. doi: 10.3389/fmicb.2014.00477. eCollection 2014. PMID 25309517
- [Background] Crimeen-Irwin B, Scalzo K, Gloster S, Mottram PL, Plebanski M. Failure of immune homeostasis -- the consequences of under and over reactivity. Curr Drug Targets Immune Endocr Metabol Disord. 2005 Dec;5(4):413-22. doi: 10.2174/156800805774912980. PMID 16375694
- [Background] Govindaraj C, Scalzo-Inguanti K, Scholzen A, Li S, Plebanski M. TNFR2 Expression on CD25(hi)FOXP3(+) T Cells Induced upon TCR Stimulation of CD4 T Cells Identifies Maximal Cytokine-Producing Effectors. Front Immunol. 2013 Aug 6;4:233. doi: 10.3389/fimmu.2013.00233. eCollection 2013. PMID 23964278
- [Background] Wilson KL, Xiang SD, Plebanski M. Montanide, Poly I:C and nanoparticle based vaccines promote differential suppressor and effector cell expansion: a study of induction of CD8 T cells to a minimal Plasmodium berghei epitope. Front Microbiol. 2015 Feb 6;6:29. doi: 10.3389/fmicb.2015.00029. eCollection 2015. PMID 25705207
- [Background] Chen X, Hamano R, Subleski JJ, Hurwitz AA, Howard OM, Oppenheim JJ. Expression of costimulatory TNFR2 induces resistance of CD4+FoxP3- conventional T cells to suppression by CD4+FoxP3+ regulatory T cells. J Immunol. 2010 Jul 1;185(1):174-82. doi: 10.4049/jimmunol.0903548. Epub 2010 Jun 4. PMID 20525892
- [Background] Flanagan KL, van Crevel R, Curtis N, Shann F, Levy O; Optimmunize Network. Heterologous ("nonspecific") and sex-differential effects of vaccines: epidemiology, clinical trials, and emerging immunologic mechanisms. Clin Infect Dis. 2013 Jul;57(2):283-9. doi: 10.1093/cid/cit209. Epub 2013 Apr 9. PMID 23572484
- [Background] Nakaya HI, Li S, Pulendran B. Systems vaccinology: learning to compute the behavior of vaccine induced immunity. Wiley Interdiscip Rev Syst Biol Med. 2012 Mar-Apr;4(2):193-205. doi: 10.1002/wsbm.163. Epub 2011 Oct 19. PMID 22012654
- [Background] Nakaya HI, Wrammert J, Lee EK, Racioppi L, Marie-Kunze S, Haining WN, Means AR, Kasturi SP, Khan N, Li GM, McCausland M, Kanchan V, Kokko KE, Li S, Elbein R, Mehta AK, Aderem A, Subbarao K, Ahmed R, Pulendran B. Systems biology of vaccination for seasonal influenza in humans. Nat Immunol. 2011 Jul 10;12(8):786-95. doi: 10.1038/ni.2067. PMID 21743478
- [Background] Furman D, Hejblum BP, Simon N, Jojic V, Dekker CL, Thiebaut R, Tibshirani RJ, Davis MM. Systems analysis of sex differences reveals an immunosuppressive role for testosterone in the response to influenza vaccination. Proc Natl Acad Sci U S A. 2014 Jan 14;111(2):869-74. doi: 10.1073/pnas.1321060111. Epub 2013 Dec 23. PMID 24367114
- [Background] Yao X, Hamilton RG, Weng NP, Xue QL, Bream JH, Li H, Tian J, Yeh SH, Resnick B, Xu X, Walston J, Fried LP, Leng SX. Frailty is associated with impairment of vaccine-induced antibody response and increase in post-vaccination influenza infection in community-dwelling older adults. Vaccine. 2011 Jul 12;29(31):5015-21. doi: 10.1016/j.vaccine.2011.04.077. Epub 2011 May 10. PMID 21565245
- [Background] Chen X, Oppenheim JJ. TNF-alpha: an activator of CD4+FoxP3+TNFR2+ regulatory T cells. Curr Dir Autoimmun. 2010;11:119-34. doi: 10.1159/000289201. Epub 2010 Feb 18. PMID 20173391
- [Background] Duraisingham SS, Rouphael N, Cavanagh MM, Nakaya HI, Goronzy JJ, Pulendran B. Systems biology of vaccination in the elderly. Curr Top Microbiol Immunol. 2013;363:117-42. doi: 10.1007/82_2012_250. PMID 22903566